CLINICAL TRIAL: NCT05004272
Title: Impact of Therapeutic Measures on Body Awareness
Brief Title: IOBA - Impact on Body Awareness
Acronym: IOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PMR_IOBA_01
Record Dates: First submitted 2021-06-02; First posted 2021-08-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Perception, Self; Body Image; Self-Assessment
MeSH Terms: interventions — Massage; Gymnastics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage (Active Comparator)
  Interventions: Procedure: Massage
- Gymnastics (Active Comparator)
  Interventions: Procedure: Gymnastics
- Lecture (Placebo Comparator)
  Interventions: Other: Lecture

INTERVENTIONS:
Procedure: Massage — 20-minute manual full-body massage
  Arms: Massage
Procedure: Gymnastics — 20-minute moderate body workout
  Arms: Gymnastics
Other: Lecture — 20-minute lecture on medicinal herbs
  Arms: Lecture

SUMMARY:
Due to social isolation and increased stress factors during the COVID-19 pandemic an increase of psychological and psychosomatic complaints in the population can be observed. There is growing evidence of the importance of body awareness (BA) in these complaints. The question arises how BA can be modified through therapeutic measures. The Awareness Body Chart (ABC), an innovative non-verbal tool for investigating subjective body awareness, implemented in clinical practice brings to light astonishing findings of patients' bodily experiences which have not been collected through verbal communication so far. In a randomized controlled study with 96 healthy adults in three groups (massage, gymnastics and control group), the use of the ABC questionnaire and further German questionnaires (Short questionnaire on self-perception of the body, self-rating mood scale - revised) concerning body awareness and well-being should analyse the following hypotheses: Primary hypothesis: There is a difference in the change of BA between the massage group and the control group, and there is a difference in the change of BA between the gymnastics group and the control group. Secondary hypothesis: There is a difference in the change of BA between the massage group and the gymnastics group. Before interventions demographic data and further questionnaires concerning health conditions of the participants (Simple Physical Activity Questionnaire, Short Form Health Survey, Brief Symptom Inventory and additional questions) are administered. Correlations between BA and the results of these tests will be investigated too. All these analyses can provide innovative information about BA and be indicative in the use of physiotherapeutic measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Signing of informed consent by participants and head of the study
* Understanding of German language in order to be able to follow a lecture and complete questionnaires

Exclusion Criteria:

* Current sick leave
* Pregnancy
* Acute physical or psychological complaints on the day of study participation
* Chronic illnesses / disabilities which make it difficult to participate in a moderate exercise while standing
* Chronic diseases / impairments that make it difficult to lie prone for a massage
* Current illnesses or injuries that are a contraindication for hand massages or gymnastics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Awareness Body Chart Questionnaire | Before intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness.
Awareness Body Chart Questionnaire | Immediately after intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness.

SECONDARY OUTCOMES:
Short questionnaire on self-perception of the body | Before intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Short questionnaire on self-perception of the body | Immediately after intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Self-rating mood scale - revised | Before intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.
Self-rating mood scale - revised | Immediately after intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.

OTHER OUTCOMES:
Simple Physical Activity Questionnaire | Before intervention
  Questionnaire to survey physical activity: It should show a snapshot of hours per day of an average day in the past week. The time in bed, the time while doing sedentary work (including dozing), while walking, while exercising and during other physical activities (such as household chores) is interrogated. The test does not measure the intensity of physical activity, but rather sorts it into the groups walking, sport and other categories.
Short Form Health Survey (SF-12) | Before intervention
  Questionnaire on health-related quality of life. It consists of twelve questions relating to the last four weeks and yields statements about eight different dimensions of subjective health: general health perception, physical health, physically-conditioned role function, physical pain, vitality, mental health, emotionally-related role function, social functionality. Different Likert-Scales are used. A physical sum scale and a psychological sum scale can be calculated. The polarity of four items must be reversed so that higher values in all items and total scales reflect a better state of health. Normative data are available.
Brief Symptom Inventory | Before intervention
  Questionnaire on the burden of symptoms. The BSI is also called the Brief Symptom Check List (BSCL), it is a short form of the SCL-90 (Derogatis, 1993). The BSI consists of 53 items (physical as well as psychological symptoms), which are assessed subjectively on a Likert scale in relation to the last seven days from 0 = "not at all" to 5 = "very strong". The items result in nine scales: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.
Body Mass Index | Before intervention
  Relation of body weight to the square of body height
Additional questions | Before intervention
  Questions on demographic data and chronic complaints and current illnesses
Charlson Comorbidity Index | Before intervention
  Questionnaire on comorbidities
Feedback form | Immediately after investigation
  Personal feedback on questionnaires and measures

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Austria